CLINICAL TRIAL: NCT00012727
Title: Matching, Outcomes and Costs in Substance Abuse/Psychiatric Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 95-011
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2005-07

CONDITIONS: Dual Diagnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Procedure: Matching Symptom Severity to Service Intensity

INTERVENTIONS:
Procedure: Matching Symptom Severity to Service Intensity

SUMMARY:
This project�s goal is to improve the quality of care and reduce treatment costs for veterans with substance abuse and psychiatric problems.

DETAILED DESCRIPTION:
Background:

This project�s goal is to improve the quality of care and reduce treatment costs for veterans with substance abuse and psychiatric problems.

Objectives:

This project is evaluating a patient-treatment matching strategy to improve residential treatment for substance abuse patients with psychiatric disorders. Its immediate objective is to examine whether the matching strategy results in more effective and cost-effective treatment in VA programs. We hypothesize that patients with severe clinical problems will have better outcomes when they are matched to service-intensive programs; patients with moderate problems will have better outcomes when they are matched to programs having a lower intensity of services. For both patient groups, community treatment should prove to be more cost-effective than hospital treatment.

Methods:

The project utilized a stratified randomized design. We paired each of three VA hospital programs that treat dual diagnosis patients and are high on intensity with a nearby high-intensity community residential facility (CRF) that contracts with the VA. We also paired four VA hospital and four CRFs that are low on intensity. Veterans who applied for substance abuse treatment at VA facilities were randomly assigned to either the VA hospital or CRF. Patient assessments have been conducted at intake (N=230), discharge, and a 4-month follow-up. Primary outcomes are patients� severity of substance abuse and psychiatric problems. Secondary outcomes are patients� functional status and their VA and non-VA health care utilization and its costs.

Status:

Completed.

ELIGIBILITY:
Inclusion Criteria:

Patients must be entering a VA inpatient substance abuse or psychiatric treatment program and be clinically judged as appropriate for inpatient or community residential care.

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Study Completion 2001-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Timko, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (6):
- United States (6):
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE, Omaha, Nebraska
  - Oklahoma City VA Medical Center, Oklahoma City, OK, Oklahoma City, Oklahoma
  - Hampton VA Medical Center, Hampton, VA, Hampton, Virginia

REFERENCES:
- [Result] Timko C, Sempel JM, Moos RH. Models of standard and intensive outpatient care in substance abuse and psychiatric treatment. Adm Policy Ment Health. 2003 May;30(5):417-36. doi: 10.1023/a:1024693614501. PMID 12940684
- [Result] Timko C, Sempel JM. Short-term outcomes of matching dual diagnosis patients' symptom severity to treatment intensity. J Subst Abuse Treat. 2004 Apr;26(3):209-18. doi: 10.1016/S0740-5472(04)00002-9. PMID 15063915
- [Result] Timko C, Lesar M, Calvi NJ, Moos RH. Trends in acute mental health care: comparing psychiatric and substance abuse treatment programs. J Behav Health Serv Res. 2003 Apr-Jun;30(2):145-60. doi: 10.1007/BF02289804. PMID 12710369
- [Result] Timko C, Lesar M, Engelbrekt M, Moos RH. Changes in services and structure in community residential treatment facilities for substance abuse patients. Psychiatr Serv. 2000 Apr;51(4):494-8. doi: 10.1176/appi.ps.51.4.494. PMID 10737825
- [Result] Timko C, Sempel JM. Intensity of acute services, self-help attendance and one-year outcomes among dual diagnosis patients. J Stud Alcohol. 2004 Mar;65(2):274-82. doi: 10.15288/jsa.2004.65.274. PMID 15151360
- [Result] Chen S, Barnett PG, Sempel JM, Timko C. Outcomes and costs of matching the intensity of dual-diagnosis treatment to patients' symptom severity. J Subst Abuse Treat. 2006 Jul;31(1):95-105. doi: 10.1016/j.jsat.2006.03.015. PMID 16814015
- [Result] Timko C, Yu K, Moos RH. Demand characteristics of residential substance abuse treatment programs. J Subst Abuse. 2000;12(4):387-403. doi: 10.1016/s0899-3289(01)00056-6. PMID 11452841